**Ketoconazole Cream 2%** 

Protocol / Study No. 71875502

#### **COVER PAGE**

#### STATISTICAL ANALYSIS PLAN

Final Version 3.0

February 28, 2019

NCT03824912

A Randomized, Double-Blind, Vehicle-Controlled, Parallel-Design, Multiple-Site Clinical Study to Evaluate the Therapeutic Equivalence of Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd) to Ketoconazole Cream 2% (G&W Laboratories Inc.) in the Treatment of Tinea Pedis

Protocol Number: 71875502

Novum Study Number: 71875502

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

#### STATISTICAL ANALYSIS PLAN

A Randomized, Double-Blind, Vehicle-Controlled, Parallel-Design, Multiple-Site Clinical Study to Evaluate the Therapeutic Equivalence of Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd) to Ketoconazole Cream 2% (G&W Laboratories Inc.) in the Treatment of Tinea Pedis

Protocol Number: 71875502 Novum Study Number: 71875502

#### **Sponsor:**

Encube Ethicals Pvt Ltd 803, B Wing, HDIL Kaledonia, Sahar Road, Andheri (E), Mumbai – 400069, Maharashtra, India

#### **Contract Research Organization:**

Novum Pharmaceutical Research Services 225 W. Station Square Drive, Suite 200 Pittsburgh, PA 15219

February 28, 2019

Final Version 3.0

**Ketoconazole Cream 2%** 

Protocol / Study No. 71875502

# SAP FINAL VERSION APPROVALS

A Randomized, Double-Blind, Vehicle-Controlled, Parallel-Design, Multiple-Site Clinical Study to Evaluate the Therapeutic Equivalence of Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd) to Ketoconazole Cream 2% (G&W Laboratories Inc.) in the Treatment of Tinea Pedis

| Written By: | |
|---|---|
| Signature: Jianhua Liu, MSc Senior Biostatistician Novum Pharmaceutical Research Services | Date: |
| Reviewed By: | |
| Signature:<br>Pina D'Angelo, MSc<br>Executive Director, Scientific Affairs (Biostatistics)<br>Novum Pharmaceutical Research Services | Date: |
| Approved By: | |
| Signature: Dr. Lalatendu Panigrahi Chief Scientific Officer Encube Ethicals Pvt Ltd | Date: |
| Approved By: | |
| Signature: Dr. Brijesh B. Wadekar Head - Clinical Trials Encube Ethicals Pvt. Ltd. | Date: |

# Ketoconazole Cream 2%

Protocol / Study No. 71875502

# **Revision History**

| VERSION | DATE | DESCRIPTION OF REVISIONS | REVISED BY |
|---|---|---|---|
| Draft 1.0 | October 4, 2018 | New Document | Jianhua Liu |
| Draft 2.0 | November 08, 2018 | Incorporate client's comments | Jianhua Liu |
| Final 1.0 | December 04, 2018 | Finalize SAP | Jianhua Liu |
| Final 2.0 | January 23, 2019 | Add missed doses to Listing L16.2.5 | Jianhua Liu |
| Final 2.0 | February 05, 2019 | Add Dr. Brijesh to the approval page | Jianhua Liu |
| Final 3.0 | February 28, 2019 | <ol> <li>To document that all subjects in the safety need to have at least one dose applied as per new guidance.</li> <li>To remove criteria of had at least one post-baseline evaluation from mITT population definition as per new guidance.</li> </ol> | Jianhua Liu |

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

#### **List of Abbreviations and Definition of Terms**

ADaM Analysis Data Model AE Adverse Event

CDISC Clinical Data Interchange Standards Consortium

CMH Cochran-Mantel-Haenszel
CRO Contract Research Organization
eCRF electronic Case Report Form
FDA Food and Drug Administration

ICF Informed Consent Form

ICH International Conference on Harmonization

IRB Institutional Review Board KOH Potassium Hydroxide

LOCF Last Observation Carried Forward

MedDRA Medical Dictionary for Regulatory Activities

mITT modified Intent-to-Treat

mL Milliliter PP Per-Protocol

SAE Serious Adverse Event
SAP Statistical Analysis Plan
SAS Statistical Analysis System
SDTM Study Data Tabulation Model
TEAE Treatment Emerget Advers Events

USA United States of America

| Ketoconazole Cream 2% Protocol / Study No. 718 | <u>75502</u> |
|---|---|
| TABLE OF CONTENTS | |
| 1. INTRODUCTION | 8 |
| 2. OBJECTIVES | |
| 3. OVERALL STUDY DESIGN | |
| 4. RANDOMIZATION AND BLINDING. | |
| 5. SAMPLE SIZE | |
| 6. EFFICACY VARIABLES AND EFFICACY ENDPOINTS | |
| 7. STUDY POPULATIONS | |
| 8. STATISTICAL ANALYSIS METHODS | |
| 8.1 Baseline Characteristics | |
| 8.1.1 Patient Disposition | |
| 8.1.2 Demographic and Other Baseline Characteristics | |
| 8.1.3 Medical History | |
| 8.2 Efficacy Analyses | |
| 8.2.1 Efficacy Analyses on Primary and Secondary Endpoints | |
| 8.3 Safety Analysis | |
| 8.3.1 Adverse Events | |
| 8.3.2 Vital Signs | 18 |
| 8.3.3 Local Signs and Symptoms | 19 |
| 8.3.4 Concomitant Medications | 19 |
| 8.4 Multiple Comparisons | 19 |
| 8.5 Methods for Handling Missing Data | |
| 8.6 Interim Analyses | 20 |
| 8.7 Changes to the Protocol Defined Statistical Analysis Plan | 20 |
| 9. TABLE, LISTING AND FIGURE SHELLS | 21 |
| T14.1.1 Summary of Patient's Disposition | 23 |
| T14.1.2 Summary of Protocol Deviations | 24 |
| T14.1.3.1 Summary of Patients Excluded from Efficacy Analysis (Randomized | |
| Population) | |
| T14.1.3.2 Summary of Patients Included in Analysis Population by Study Site | |
| T14.2.1 Summary of Demographic Data (Safety Population) | 28 |
| T14.2.2 Summary of Baseline Characteristics (Safety Population) | |
| T14.2.3 Summary of Demographic Data (modified Intent-to-Treat Population) | 33 |
| T14.2.4 Summary of Baseline Characteristics (modified Intent-to-Treat Population) | 33 |
| T14.2.5 Summary of Demographic Data (Per-Protocol Population) | |
| T14.2.6 Summary of Baseline Characteristics (Per-Protocol Population) | 33 |
| T14.2.7.1 Summary of Total Severity Score of Local Signs and Symptoms (modified | |
| Intent-to-Treat Population) | 34 |
| T14.2.7.2 Summary of Total Severity Score of Local Signs and Symptoms (Per- | |
| Protocol Population) | 34 |
| T14.2.8.1 Summary of KOH Wet Mount and Mycological Culture (modified Intent- | |
| to-Treat Population) | 35 |

| Ketoconazole Cream 2% | Protocol / Study No. 71875502 |
|---|---|
| T14.2.8.2 Summary of KOH Wet Mount and Mycological | |
| Population) | |
| T14.2.9 Summary of Analysis Results of Primary Efficacy<br>Patients in each Treatment Group with a Therapeutic | Cure of Tinea Pedis at the |
| Test-of-cure Visit (Day $56 \pm 4$ ) | 36 |
| T14.2.10 Summary of Analysis Results of Secondary Efficients in each Treatment Group Who are Considere | d a Clinical Cure at Day 56 |
| ± 4 | cacy Endpoint Proportion of d a Mycological Cure at Day |
| $56 \pm 4$ | 38 |
| T14.3.1 Overall Summary of Adverse Events (Safety Pop | |
| T14.3.2 Summary of Frequency of Adverse Events by Boo Population) | ` ' |
| T14.3.3 Summary of Frequency of Adverse Events by Rel Population) | ationship (Safety |
| T14.3.4 Summary of Frequency of Adverse Events by Sev | |
| T14.3.5 Summary of Frequency of Serious Adverse Event | |
| T14.3.6 Summary of Vital Signs (Safety Population) | · • • • · |
| L16.2.1 Listing of Discontinued Patients | |
| L16.2.2 Listing of Protocol Deviations | |
| L16.2.3.1 Listing of Patients Excluded from the Per-Proto | |
| L16.2.3.2 Listing of Patients Excluded from the modified | * |
| L16.2.4.1 Listing of Demographic Data | |
| L16.2.4.2 Listing of Medical History | |
| L16.2.4.3 Listing of Prior and Concomitant Medication | |
| L16.2.5 Listing of Drug Administration | 51 |
| L16.2.6.1 Listing of Local Signs and Symptoms | |
| L16.2.6.2 Listing of Mycological Culture and KOH Wet N | |
| L16.2.7.1 Listing of Treatment Emergent Adverse Events | |
| L16.2.7.2 Listing of Pre-treatment Adverse Events | |
| L16.2.8.1 Listing of Pregnancy Test Results | |
| L16.2.8.2 Listing of Vital Signs | |

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

#### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) is based on the final Clinical Study Protocol 71875502 (Novum Study No. 71875502) Rev. 0 dated 06/13/2018. The SAP provides details on the planned statistical methodology for the analysis of the study data. The SAP also outlines the statistical programming specifications for the tables, listings and figures.

This SAP describes the study endpoints, derived variables, anticipated data transformations and manipulations, and other details of the analyses not provided in the study protocol. This SAP therefore outlines in detail all other aspects pertaining to the planned analyses and presentations for this study.

The following documents were reviewed in preparation of this SAP:

- Final Clinical Study Protocol 71875502 (Novum Study No. 71875502) Rev. 0 dated 06/13/2018
- Casebook for Novum Study No. 71875502

The reader of this SAP is encouraged to also read the clinical protocol for details on the conduct of this study, and the operational aspects of clinical assessments and timing for completing a patient in this study.

#### 2. OBJECTIVES

- 1. Evaluate the therapeutic equivalence of a generic Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd) to the Reference product, Ketoconazole Cream 2% (G&W Laboratories Inc.) in the treatment of tinea pedis.
- 2. Demonstrate the superiority of the clinical effect of the Test and Reference (active) products over that of the Placebo (vehicle) in the treatment of tinea pedis.
- 3. Compare the safety of the Test, Reference and Placebo products in the treatment of tinea pedis.

#### 3. OVERALL STUDY DESIGN

This randomized, double-blind, vehicle-controlled, parallel-group, multiple-site study has been designed to evaluate the clinical (therapeutic) effect of a generic Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd) compared to the Orange Book Reference Standard (RS) product, Ketoconazole Cream 2% (G&W Laboratories Inc.) in patients with tinea pedis. Additionally, both the Test and Reference (i.e., the RS) treatments will be tested for superiority to a Placebo.

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

Before any study-specific procedures are performed, all patients will read and sign the IRB-approved informed consent form (ICF).

Approximately 830 eligible patients, 18 years of age and older, will be randomized in a 2:2:1 ratio (Test: Reference: Placebo) to one of the three study products as follows:

- **Test**: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)
- **Reference**: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.))
- Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

Patients will complete three clinic visits as follows:

- Visit 1 (Day 1): Screening/Baseline
- Visit 2 (Day  $42 \pm 4$ ): End of Treatment
- Visit 3 (Day  $56 \pm 4$ ): Test-of-Cure/End of Study

Patients will be instructed to apply the study product to affected and immediate surrounding areas once daily for a total of  $42 \pm 4$  days starting on the day of enrollment (i.e., Day 1). The last dose should be applied on the day of Visit 2 (Day  $42 \pm 4$ ). Evaluations will be performed in accordance with the study schematic. Safety assessments will include monitoring of adverse events (AEs), vital signs measurement, and urine pregnancy tests (for females of childbearing potential). Clinical assessments will include the potassium hydroxide (KOH) wet mount, mycological culture, and rating of signs and symptoms. The Investigator should identify the most severe lesion (i.e., target lesion) at baseline. Although the study product should be applied to all infected areas (both feet), only the target lesion will be evaluated for analysis.

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

**Figure 1 Study Schematic** 

| PROCEDURE | VISIT 1<br>(Day 1)<br>Screening/<br>Baseline | VISIT 2 (Day 42 ± 4 Days)* End of Treatment | VISIT 3<br>(Day 56 ± 4 Days)<br>Test-of-Cure/<br>End of Study |
|---|---|---|---|
| Informed Consent | X | | |
| Medical History and<br>Demographics | X | | |
| Perform Pregnancy Test** | X | X | X |
| Record Vital Signs | X | X | X |
| Review and Assessment of<br>Concomitant Medications | X | X | X |
| Review and Assessment of<br>Adverse Events | | X | X |
| Designate Target Lesion | X | | |
| Assess Local Signs and<br>Symptoms | X | X | X |
| Collect Sample for KOH Wet<br>Mount | X | | $\chi^{\dagger}$ |
| Inclusion/Exclusion Criteria<br>Review | X | | |
| Collect Sample for Mycological Culture <sup>‡</sup> | X | | X |
| Dispense Study Product | X | | |
| Provide Patient Diary | X | X | |
| Collect/Review Patient Diary | | X | X |
| Collect Study Product | | X | $X^{\S}$ |
| Discharge from Study | 42 4 1 | 41 - 1 6 11 | X |

<sup>\*</sup>Dosing regimen is once daily for  $42 \pm 4$  days starting on the day of enrollment (Day 1) through the day of Visit 2 (Day  $42 \pm 4$ ).

<sup>\*\*</sup>For females of childbearing potential

<sup>&</sup>lt;sup>†</sup>KOH sample will not be collected if baseline culture is negative.

<sup>&</sup>lt;sup>‡</sup>Mycological culture sample will not be sent if KOH is negative at baseline or positive at Visit 3. See Appendix B.

<sup>§</sup>Study product will be collected at Visit 3 if it is not returned at Visit 2.

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

#### 4. RANDOMIZATION AND BLINDING

All randomized study product will be blinded and packaged in sealed boxes by an independent packaging company. Randomization will be pre-planned according to a computer-generated randomization schedule. The randomization will be generated in blocks, each containing five patients' worth of study product (2 Test, 2 Reference, and 1 Placebo).

The randomization/patient number will be a unique four-digit number. This number will be assigned immediately before dispensing of study product and in ascending sequential order, beginning with the lowest available number at the study site. Each patient kit and each dispensed study tube should include the four-digit patient number on the label.

At the end of the study, after all the clinical data have been entered and the study database has been locked, a copy of the randomization schedule will be sent to the statistician.

The Investigator, staff at the study site, study monitors, and data analysis/management personnel will be blinded to the patient assignment.

#### 5. SAMPLE SIZE

For the primary endpoint analysis (proportion of patients in the PP population with a Therapeutic Cure at the test-of-cure visit), sample size is estimated for therapeutic equivalence of the Test to the Reference product and superiority of each of the active treatments groups over Placebo. The sample size estimations are based on previous studies conducted for ketoconazole cream (Teva Pharmaceuticals; ANDA 75-581). Readers are encouraged to see the protocol reference list for the results of the previous studies used for sample size calculation.

In the PP population, the proportion of patients with a Therapeutic Cure in the Reference group is expected to be 50%. Assuming that the Therapeutic Cure rate for the Test treatment group is an absolute difference of 5% lower than the Reference Responder rate (i.e.,  $p_T$  -  $p_R$  = -5%), a sample size of 172 patients in each active group in the PP population will provide approximately 85% power to demonstrate therapeutic equivalence (i.e., the 90% confidence interval [Yates' continuity-corrected] on the  $p_T$  -  $p_R$  difference is within a defined equivalence range [-20%, +20%]).

The Therapeutic Cure rates for the Placebo and active treatment groups at the test-of-cure visit are anticipated to be approximately 10% and at least 40% (Test = 40%, Reference = 45%), respectively, in the mITT population. Using a 2:1 (Active: Placebo) randomization scheme, and assuming the conversion rate from mITT to PP will be approximately 80%, 216 patients in each active treatment group (Test and Reference) and 108 patients in the Placebo group of the mITT population will provide at least 99% power to demonstrate superiority of active treatments over Placebo (p < 0.05; using two-sided, continuity-corrected Z-test and a pooled response rate for the standard error of the difference in proportions).

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

Under the above assumptions, the overall study power to demonstrate therapeutic equivalence and superiority is estimated to be at least 85% ( $100\% \times 0.85 \times 0.999$ ), assuming 100% correlation between the two superiority tests.

To allow for approximately 35% of patients who may have negative fungal cultures post-randomization, drop out from the study or are otherwise non-evaluable, approximately 830 patients may be randomized (332 in each active group and 166 in the Placebo group) to yield 540 patients in the mITT population.

More than 50% of the patients should have baseline fungal cultures that test positive for T.rubrum. If fewer than 50% of enrolled patients have a positive T.rubrum culture or the number of patients with negative fungal cultures is more than anticipated, then additional patients may be enrolled to ensure that at least 430 (172:172:86) patients are eligible in the PP population, of which > 50% have a positive T.rubrum culture at baseline.

#### 6. EFFICACY VARIABLES AND EFFICACY ENDPOINTS

# **Efficacy Variables**

The primary and secondary efficacy variables are the outcome of the KOH test (negative or positive), outcome of the mycological culture (negative or positive), and signs and symptoms scores.

#### **Primary Efficacy Endpoint:**

The primary efficacy endpoint is the proportion of patients in each treatment group with a Therapeutic Cure of tinea pedis at the test-of-cure visit two weeks after the end of treatment (Day  $56 \pm 4$ ).

#### **Secondary Efficacy Endpoints:**

The secondary efficacy endpoints are:

- The proportion of patients in each treatment group with a Clinical Cure at Day  $56 \pm 4$ .
- The proportion of patients in each treatment group with a Mycological Cure at Day  $56 \pm 4$ .

#### **Definitions**

- 1. <u>Therapeutic Cure:</u> To be considered a Therapeutic Cure, the patient must have both Clinical and Mycological Cure of tinea pedis.
- 2. Therapeutic Failure: A patient will be considered a Therapeutic Failure if:

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

- a. the patient is a Clinical or Mycological Failure
- b. the patient was considered to have an insufficient therapeutic response
- c. the patient used topical drug therapy for irritation or pruritus on the feet between Visit 2 (Day  $42 \pm 4$  days) and Visit 3 (Day  $56 \pm 4$  days)
- 3. <u>Clinical Cure:</u> To be considered a clinical cure the patient's total severity score must be ≤ 2 with no individual severity score > 1.
- 4. <u>Clinical Failure:</u> A patient will be considered a Clinical Failure if the patient's total severity score is > 2 <u>or</u> any individual score is > 1.
- 5. <u>Mycological Cure:</u> To be considered a mycological cure the patient must have a negative KOH test <u>and</u> a negative fungal culture.
- 6. <u>Mycological Failure:</u> A patient will be considered a Mycological Failure if the patient's KOH test is positive <u>or</u> the patient's fungal culture is positive.

#### 7. STUDY POPULATIONS

#### **Per-Protocol Population**

The PP population will include all randomized patients who:

- Met all inclusion and exclusion criteria.
- Made the final study visit within the protocol window of Day  $56 \pm 4$  days (Day 52 to Day 60 inclusive) with no protocol violations that would affect the treatment evaluation.
- Did not have any significant protocol deviations.
- Were compliant with dosing between 75%-125% of the required doses.
- Had a positive baseline KOH and fungal culture for *Trichophyton rubrum*, *Trichophyton mentagrophyties* or *Epidermophyton floccosum*.

Patients discontinued from the study because of lack of treatment effect after completing at least 14 days of treatment will be included in the PP population as Therapeutic Failures provided they had a positive baseline KOH, positive baseline fungal culture, and did not have any significant protocol deviations. For these patients, there will be no mycological testing at time of discontinuation; therefore, they will be considered Therapeutic Failures in the primary analysis but the Mycological Cure data will be set to missing for the secondary endpoint.

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

Patients who meet the criteria above, but who also used topical drug therapy for irritation or pruritus on the feet after the treatment phase of the study will be included in the PP population as Therapeutic Failures. If no mycological testing is performed, the patients will be considered Therapeutic Failures in the primary analysis but the Mycological Cure data will be set to missing for the secondary endpoint.

All analyses performed using the PP population will be done on an observed case basis (i.e., no last observation carried forward [LOCF] will be performed).

#### **Modified Intent-to-Treat Population**

The mITT population will include randomized patients who:

- Met all inclusion/exclusion criteria.
- Applied at least one dose of assigned product.
- Had a positive baseline KOH and fungal culture for *Trichophyton rubrum*, *Trichophyton mentagrophyties* or *Epidermophyton floccosum*.

Patients discontinued early for reasons other than lack of treatment effect will be excluded from the PP population and included in the mITT population using LOCF. Patients who qualify for inclusion in the mITT population with missing endpoint data who were not discontinued for lack of treatment effect will also be evaluated using LOCF; that is, if a patient who was not discontinued for lack of treatment effect does not have KOH or mycological culture results at Visit 3, this patient will be evaluated for the primary and secondary endpoints using LOCF from Visit 1. Patients who discontinued because of lack of treatment effect will not have LOCF performed.

Patients who meet the criteria above, but who also used topical drug therapy on the feet for the treatment of irritation or pruritus after the treatment phase of the study will be included in the mITT as Therapeutic Failures. If no mycological testing is performed, these patients will be considered Therapeutic Failures in the primary analysis but the Mycological Cure data will be set to missing for the secondary endpoint. No LOCF will be performed.

#### **Safety Population**

The Safety population will include all randomized patients who use at least one dose of product.

#### 8. STATISTICAL ANALYSIS METHODS

If not otherwise specified, statistical significance is defined as p < 0.05 and is two-tailed. Data will be summarized with respect to demographic and baseline characteristics and safety

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

variables.

For categorical variables, the number and percent of each category within a parameter will be calculated. For continuous variables, statistics will include n, mean, standard deviation, median and range.

All statistical analyses will be conducted using SAS®, Version 9.4 or higher. Datasets will be prepared using headings from Clinical Data Interchange Consortium (CDISC) Study Data Tabulation Model (SDTM) implementation for human clinical trials and ADaM (Analysis Dataset Model) and FDA Guidance of Technical Specifications - Comparative Clinical Endpoints Bioequivalence Study Analysis Datasets for Abbreviated New Drug Application (September 2018).

#### 8.1 Baseline Characteristics

#### **8.1.1 Patient Disposition**

The patient disposition information will be summarized by treatment group as well as total. The number of patients randomized will be tabulated by treatment group and total. In addition, completion status and primary reason for withdrawal will be summarized by treatment group and total.

#### 8.1.2 Demographic and Other Baseline Characteristics

Baseline comparability of all treatment groups will be evaluated separately in the PP, mITT and Safety populations.

The following baseline demographics (determined from their initial study visit) will be evaluated:

- Age (years)
- Sex (male/female)
- Ethnicity (Hispanic/non-Hispanic)
- Race (White, Black/African American, Native Hawaiian or Other Pacific Islander, Asian, American Indian or Alaska Native, Other)
- Type of infection (interdigital only or interdigital with extension)
- Total baseline signs and symptoms score
- Presence or absence of onychomycosis
- Number of Tinea Pedis infections in the past 12 months

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

#### • Primary infective organism

Summary tables by treatment group will be presented. Continuous variables will be summarized using descriptive statistics (n, mean, standard deviation, median and range). Range will have the same decimal places as raw values. Mean, median and standard deviation will have one decimal place more than that of raw values. Categorical variables will be summarized using frequencies and percentage.

Baseline comparability of the treatments will be presented using Cochran-Mantel-Haenszel (CMH) test for the categorical variables, and Analysis of Variance for the continuous variables.

All data will be listed by treatment group and patient.

#### **8.1.3 Medical History**

At Visit 1, Patients will also be questioned about personal medical history, including tinea pedis history.

Medical history data will be listed by treatment group and patient.

# **8.2 Efficacy Analyses**

#### 8.2.1 Efficacy Analyses on Primary and Secondary Endpoints

#### Therapeutic Equivalence

Therapeutic equivalence will be evaluated for the primary endpoint in the per-protocol (PP) population. If the 90% confidence interval (calculated using Yates' continuity correction) on the absolute difference between the proportion of patients with a Therapeutic Cure in the Test and Reference groups  $(p_T - p_R)$  is contained within the range [-20%, +20%] then therapeutic equivalence of the Test product to the Reference product will be considered to have been demonstrated.

The same statistical approach will be conducted for analyses of the secondary endpoints in the PP population.

To declare therapeutic equivalence of the Test product to the Reference product, equivalence must be demonstrated for only the primary endpoint in the PP population.

Patients who are missing mycological culture data at the test-of-cure visit will not be included in the analysis for the secondary endpoint of Mycological Cure.

#### Superiority to Placebo

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

Superiority of the Test and Reference products against the Placebo product for the primary endpoint will be evaluated in the mITT population using, if necessary, LOCF as described in section 11.3.2 of the protocol.

Patients discontinued early for reasons other than lack of treatment effect will be excluded from the PP population and included in the mITT population using LOCF. Patients who qualify for inclusion in the mITT population with missing endpoint data who were not discontinued for lack of treatment effect will also be evaluated using LOCF; that is, if a patient who was not discontinued for lack of treatment effect does not have KOH or mycological culture results at Visit 3, this patient will be evaluated for the primary and secondary endpoints using LOCF from Visit 1. Patients who discontinued because of lack of treatment will not have LOCF performed.

Patients who meet the criteria above, but who also used topical drug therapy on the feet for the treatment of irritation or pruritus after the treatment phase of the study will be included in the mITT as Therapeutic Failures. If no mycological testing is performed, these patients will be considered Therapeutic Failures in the primary analysis but the Mycological Cure data will be set to missing for the secondary endpoint. No LOCF will be performed.

If the proportions of patients with a Therapeutic Cure in the Test and the Reference product groups are numerically and statistically superior to that of the Placebo (p < 0.05; using a two-sided Cochran-Mantel-Haenszel [CMH] test, stratified by clinical site) then superiority of the Test and Reference products over Placebo will be concluded.

The same statistical approach will be conducted for analyses of the secondary endpoints in the mITT population.

To declare superiority of the Test and Reference products over Placebo, their superiority must be demonstrated for only the primary endpoint in the mITT population.

#### Treatment-by-Site Interaction and Pooling of Clinical Sites

As this is a multiple-site study, the interaction of treatment-by-site may be evaluated for the primary efficacy endpoint in the PP population for equivalence testing. The treatment-by-site interaction will be evaluated by the Breslow-Day test for homogeneity of the odds ratio at the 5% significance level (p < 0.05, 2-sided). A site(s) with a low enrollment rate(s) may be pooled with its geographically closest site, so as to avoid bias in the stratification of the sites in the CMH test and in the estimation of a treatment-by-site interaction effect. The pooling will be done for low enrolling sites that account for less than 4-7% of the total number of patients in the PP population at the site with the highest enrolling rate in the PP population. If the treatment-by-site interaction term is found to be statistically significant (p < 0.05) for the primary endpoint, then the interaction term will also be assessed for clinical relevance before pooling the data across sites. This will include examination of Therapeutic Cure rates at each site where sample sizes per treatment may be influential in the assessment of the interaction. The treatment-by-site

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

interaction may also be evaluated for the analyses of the secondary endpoints in the PP population for equivalence testing if the treatment-by-site interaction is found to be significant in the primary analysis.

#### 8.3 Safety Analysis

#### **8.3.1** Adverse Events

All the adverse events (AEs) reported throughout the study will be coded and classified according to the MedDRA (Medical Dictionary for Regulatory Activities) coding dictionary (Version 21.0 or higher).

Treatment emergent adverse events (TEAE) are those that have a start date after the study treatment has been administered or the events that were present before administration of study treatment and worsen in severity after administration of study treatment. Treatment emergent adverse events will be summarized and analyzed in a summary table. Pre-treatment adverse events will be presented in the listing.

A summary table of the number and percent of patients with TEAEs by system organ class, preferred term, and treatment will be presented. Each patient will be counted only once within each preferred term.

A frequency summary table of the number of TEAEs by system organ class, preferred term, severity, and treatment will be presented. Severity will be classified as "Mild", "Moderate", or "Severe".

Similarly, a frequency summary table of the number of TEAEs by system organ class, preferred term, and relationship to a study drug, and treatment will be presented. Relationship to a study drug will be classified as "Not Related" or "Related".

If sufficient data exist, then TEAE frequencies will be compared among the three treatments using Fisher's exact test; if this test is statistically significant at the 5% significance level, then a pairwise Fisher's exact test comparing Test and Reference will be conducted.

TEAEs will be listed by treatment group and patient. Pre-treatment adverse events will be listed by patient.

#### 8.3.2 Vital Signs

The patient's vital signs will be recorded (pulse, blood pressure, temperature and respiration rate) at each visit.

Descriptive summaries (number of observations, mean, standard deviation, minimum, median and maximum) will be provided by treatment group and visit.

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

#### 8.3.3 Local Signs and Symptoms

The Clinical Signs and Symptoms of tinea pedis will be rated by the Investigator as "none", "mild," "moderate" or "severe" using the following standardized rating scale.

- 0 =None (complete absence of any sign or symptom)
- 1 = Mild (Slight)
- 2 = Moderate (Definitely Present)
- 3 = Severe (Marked, Intense)

The following signs and symptoms will be rated at each visit:

- Signs: Fissuring/cracking, erythema, maceration, and scaling
- Symptoms: Pruritus and burning/stinging

A frequency summary table comparing the signs and symptoms for each treatment group will be presented by visit.

All data will be listed by treatment group and patient.

#### **8.3.4 Concomitant Medications**

At Visit 1, patients will be questioned about medication use over the previous six months. At all subsequent visits, patients will be questioned about ongoing or new concomitant medication use.

All prior and concomitant medications taken since screening until the end of the study will be listed by treatment group and patient.

#### **8.4 Multiple Comparisons**

No multiple comparison adjustment will be made in this study.

#### 8.5 Methods for Handling Missing Data

For demographic and baseline characteristics, each variable will be analyzed using all available data. Patients with missing data will be excluded only from analyses for which data are not available

Superiority of the Test and Reference products against the Placebo product for the primary endpoint will be evaluated in the mITT population using LOCF.

Patients discontinued early for reasons other than lack of treatment effect will be excluded from the PP population and included in the mITT population using LOCF. Patients who qualify for inclusion in the mITT population with missing endpoint data who were not discontinued for lack

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

of treatment effect will also be evaluated using LOCF; that is, if a patient who was not discontinued for lack of treatment effect does not have KOH or mycological culture results at Visit 3, this patient will be evaluated for the primary and secondary endpoints using LOCF from Visit 1. Patients who discontinued because of lack of treatment will not have LOCF performed.

Patients who meet the criteria above, but who also used topical drug therapy on the feet for the treatment of irritation or pruritus after the treatment phase of the study will be included in the mITT as Therapeutic Failures. If no mycological testing is performed, these patients will be considered Therapeutic Failures in the primary analysis but the Mycological Cure data will be set to missing for the secondary endpoint. No LOCF will be performed.

# **8.6 Interim Analyses**

There is no interim analysis planned in this study.

#### 8.7 Changes to the Protocol Defined Statistical Analysis Plan

To conform to recommendations in the recently updated Draft Guidance on Ketoconazole (Revised Feb 2019), the following changes to the statistical analyses described in the protocol will be made.

| Wordings in protocol | Changed to |
|---|---|
| Protocol section 11.3.3 The Safety population will include all patients who are randomized and received study product. | The Safety population will include all randomized patients who use at least one dose of product. |
| Protocol section 11.3.2 The mITT population will include randomized patients who: • Met all inclusion/exclusion criteria. • Applied at least one dose of assigned product. • Had at least one post-baseline evaluation. • Had a positive baseline KOH and fungal culture for <i>Trichophyton rubrum</i> , <i>Trichophyton mentagrophyties</i> or <i>Epidermophyton floccosum</i> . | The mITT population will include randomized patients who: • Met all inclusion/exclusion criteria. • Applied at least one dose of assigned product. • Had a positive baseline KOH and fungal culture for Trichophyton rubrum, Trichophyton mentagrophyties or Epidermophyton floccosum. |

**Ketoconazole Cream 2%** 

Protocol / Study No. 71875502

# 9. TABLE, LISTING AND FIGURE SHELLS

The following shells provide a framework for the display of data from this study. These shells may not be reflective of every aspect of this study but are intended to show the general layout of the Tables, Listings and Figures that will be included in the final clinical study report. Tables, Listings and Figures are numbered following the ICH structure. Table headers, variables names and footnotes will be modified as needed following data analyses. All descriptive and inferential statistical analyses will be performed using SAS® statistical software Version 9.4 or higher, unless otherwise noted.

**Ketoconazole Cream 2%** 

Protocol / Study No. 71875502

TABLE, LISTING AND FIGURE SHELLS

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

# **T14.1.1 Summary of Patient's Disposition**

# (Randomized Population)

| Patients Randomized | Test<br>N = xxx<br>n (%) | Reference<br>N = xxx<br>n (%) | Placebo<br>N = xxx<br>n (%) | Total<br>N = xxx<br>n (%) |
|---|---|---|---|---|
| Completed Study | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Terminated Early | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Adverse event | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Lack of efficacy | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Lost to follow-up | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Negative baseline culture result | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Noncompliance with study drug | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Patient scheduled/came in early for Visit 3 | | | | |
| Pregnancy | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Protocol deviation | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Significant worsening of condition requiring alternative or supplemental therapy | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Withdrawal by subject | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx(xx.x) |
| Other | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

N = number of patients randomized in that particular group; n = number of patients with data available for that particular group; total % is based on N

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX Page 1 of N

**Ketoconazole Cream 2%** 

Protocol / Study No. 71875502

# **T14.1.2 Summary of Protocol Deviations**

# (Randomized Population)

| Patients Randomized | Test<br>N = xxx<br>n (%) | Reference<br>N = xxx<br>n (%) | Placebo<br>N = xxx<br>n (%) | Total<br>N = xxx<br>n (%) |
|---|---|---|---|---|
| Total Patients with Protocol Deviations | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Total Deviations | XXX | XXX | XXX | XXX |
| Lost to follow-up | xxx | XXX | XXX | XXX |
| Missed visit | XXX | XXX | XXX | XXX |
| Noncompliance with study product | XXX | XXX | XXX | XXX |
| Noncompliance with study procedures | XXX | XXX | XXX | XXX |
| Outside visit window | XXX | XXX | XXX | XXX |
| Randomized in error | XXX | XXX | XXX | XXX |
| Restricted medication | XXX | XXX | xxx | XXX |
| Other | XXX | XXX | XXX | XXX |

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

N = number of patients randomized in that particular group; n = number of patients with data available for that particular group; total % is based on N

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX

**Ketoconazole Cream 2%** 

Protocol / Study No. 71875502

T14.1.3.1 Summary of Patients Excluded from Efficacy Analysis (Randomized Population)

| | Test<br>N = xxx<br>n (%) | Reference<br>N = xxx<br>n (%) | Placebo<br>N = xxx<br>n (%) | Total<br>N = xxx<br>n (%) |
|---|---|---|---|---|
| Safety Population | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Excluded from Safety population | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Did not receive study product | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| mITT Population | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Excluded from mITT population | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Inclusion/Exclusion criteria not met | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Did not have at least one post-baseline evaluation | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Etc. | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| PP Population | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Excluded from PP population | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Significant protocol deviations | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Etc. | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

N = number of patients randomized in that particular group; n = number of patients with data available for that particular group; total % is based on N

Programming note: exclusion reasons are not duplicated across the populations.

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX

# T14.1.3.2 Summary of Patients Included in Analysis Population by Study Site

# (Randomized population)

| | | | | 1 | Safety | | | | mITT | | | | PP | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Site<br>No. | Name | Total<br>Randomized | Test | Ref | Placebo | Total | Test | Ref | Placebo | Total | Test | Ref | Placebo | Total |
| XX | XXXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XX | XXXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

■ Encube Ethicals Pvt Ltd ■

# **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

# **T14.1.3.3 Study Timelines (Randomized Patients)**

| | Trial Timelines |
|---|---|
| | Date |
| First Patient First Visit (FPFV) | mm/dd/yyyy |
| ast Patient Last Visit (LPLV) | mm/dd/yyyy |
| rial Duration (Days) | XXX |
| Note: Trial Duration (Days) = (Date of LPLV - Date of FPFV) + 1 | |

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX

**Ketoconazole Cream 2%** 

Protocol / Study No. 71875502

T14.2.1 Summary of Demographic Data (Safety Population)

| | | Test<br>(N = xxx)<br>n (%) | Reference<br>(N = xxx)<br>n (%) | Placebo<br>(N = xxx)<br>n (%) | P-value |
|---|---|---|---|---|---|
| Age (years) | n | XXX | XXX | XXX | x.xxxx |
| | $Mean \pm SD$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | |
| | Median | XX.X | XX.X | XX.X | |
| | Range | xx-xx | xx-xx | xx-xx | |
| Age Groups | < 18 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | x.xxxx |
| | 18 - 40 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |
| | 41 - 64 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |
| | 65 – 75 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |
| | > 75 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |
| Race | American Indian or Alaska Native | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | x.xxxx |
| | Asian | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |
| | Black/African American | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |
| | Native Hawaiian or other Pacific Islander | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |
| | White | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |
| | Multiple | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

N = number of patients in the Safety Population in that particular group; n = number of patients with data available for that particular group; total % is based on N

P-values are from Cochran-Mantel-Haenszel (CMH) test for the categorical variables, and Analysis of Variance for the continuous variables.

**Ketoconazole Cream 2%** Protocol / Study No. 71875502

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX Created on: ddmmmyy hh:mm Page 1 of N

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX

# T14.2.1 Summary of Demographic Data (Safety Population)

| | | Test<br>(N = xxx)<br>n (%) | Reference<br>(N = xxx)<br>n (%) | Placebo<br>(N = xxx)<br>n (%) | P-value |
|---|---|---|---|---|---|
| Sex | Male | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | x.xxxx |
| | Female | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |
| Ethnicity | Hispanic or Latino | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | x.xxxx |
| | Not Hispanic or Latino | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

N = number of patients in the Safety Population in that particular group; n = number of patients with data available for that particular group; total % is based on N

P-values are from Cochran-Mantel-Haenszel (CMH) test for the categorical variables, and Analysis of Variance for the continuous variables.

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

T14.2.2 Summary of Baseline Characteristics (Safety Population)

| | | Test (N = xxx) | Reference<br>(N = xxx) | $ \begin{array}{l} Placebo \\ (N = xxx) \end{array} $ | Overall<br>P-value | P-value<br>Test vs.<br>Reference |
|---|---|---|---|---|---|---|
| Type of infection, n (%) | Interdigital | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | x.xxxx | X.XXXX |
| | Interdigital with extension | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | | |
| Onychomycosis, n (%) | Presence | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | X.XXXX | X.XXXX |
| | Absence | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | | |
| Primary infective organism, 1 (%) | xxxxx | xxx (x.x) | xxx (xx.x) | xxx (xx.x) | | x.xxxx |
| | XXXXX | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | | |
| Fotal baseline signs and symptom score, n (%) | n | XXX | xxx | xxx | X.XXXX | x.xxxx |
| | $Mean \pm SD$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | | |
| | Median | XX.X | XX.X | XX.X | | |
| | Range | xx-xx | xx-xx | xx-xx | | |
| Number of Tinea Pedis infections in the past 12 months, n (%) | n | xxx | xxx | XXX | x.xxxx | x.xxxx |
| | $Mean \pm SD$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | | |
| | Median | XX.X | XX.X | XX.X | | |
| | Range | xx-xx | xx-xx | xx-xx | | |

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

N = number of patients in the Safety Population in that particular group; n = number of patients with data available for that particular group; total % is based on N

**Ketoconazole Cream 2%** 

Protocol / Study No. 71875502

P-values are from Cochran-Mantel-Haenszel (CMH) test for the categorical variables, and Analysis of Variance for the continuous variables.

Note to programmer: If the overall P-value is statistically significant among the three treatment groups at the 5% alpha level (i.e. p < 0.05), then ANOVA or CMH test using only the test and reference groups will be performed to identify any potential statistically significant differences that are clinically relevant between the two active treatment groups.

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX

**Ketoconazole Cream 2%** 

Protocol / Study No. 71875502

Similar tables will be created for T14.2.3, T14.2.4, T14.2.5 and T14.2.6

T14.2.3 Summary of Demographic Data (modified Intent-to-Treat Population)

T14.2.4 Summary of Baseline Characteristics (modified Intent-to-Treat Population)

T14.2.5 Summary of Demographic Data (Per-Protocol Population)

T14.2.6 Summary of Baseline Characteristics (Per-Protocol Population)

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

T14.2.7.1 Summary of Total Severity Score of Local Signs and Symptoms (modified Intent-to-Treat Population)

| Visit | Total<br>Severity Score | Test<br>N = xxx<br>n (%) | Reference<br>N = xxx<br>n (%) | Placebo<br>N = xxx<br>n (%) |
|---|---|---|---|---|
| 1 | <=2 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | >2 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| 2 | <=2 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | >2 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| 3/Early termination | <=2 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| · | >2 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX


Similar table will be created for:

T14.2.7.2 Summary of Total Severity Score of Local Signs and Symptoms (Per-Protocol Population)

**Ketoconazole Cream 2%** 

Protocol / Study No. 71875502

T14.2.8.1 Summary of KOH Wet Mount and Mycological Culture (modified Intent-to-Treat Population)

| | ¥7* */ | D 1/ | Test | Reference | Placebo |
|---|---|---|---|---|---|
| | Visit | Result | N = xxx | N = xxx | N = xxx |
| | | | n (%) | n (%) | n (%) |
| KOH Wet Mount | 1 | Positive | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) |
| | | Negative | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) |
| | 2 | Positive | xxx(xx.x) | xxx (xx.x) | xxx (xx.x) |
| | | Negative | xxx(xx.x) | xxx (xx.x) | xxx (xx.x) |
| | 3/Early termination | Positive | xxx(xx.x) | xxx (xx.x) | xxx (xx.x) |
| | - | Negative | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Mycological Culture | 1 | Positive | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | | Negative | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | 2 | Positive | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | | Negative | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | 3/Early termination | Positive | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | • | Negative | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX


Similar table will be created for:

T14.2.8.2 Summary of KOH Wet Mount and Mycological Culture (Per-Protocol Population)

**Ketoconazole Cream 2%** 

Protocol / Study No. 71875502

# T14.2.9 Summary of Analysis Results of Primary Efficacy Endpoint Proportion of Patients in each Treatment Group with a Therapeutic Cure of Tinea Pedis at the Test-of-cure Visit (Day $56 \pm 4$ )

| Equivalence: Per-Protocol Population | | | | | |
|---|---|---|---|---|---|
| | | | _ | Difference Between Treatments | |
| Treatment<br>Group | Number of Patients (N) | Number of Patients with<br>Therapeutic Cure (n) | Proportion of Therapeutic Cure (%) | Difference (%) | 90% CI Evaluation |
| Test | XXX | XXX | XX.X | | |
| Reference | xxx | xxx | xx.x | XX.X | xx.x - xx.x |

# **Superiority: modified Intent-to-Treat Population**

| | | | _ | Treatment v | s. Placebo |
|---|---|---|---|---|---|
| Treatment<br>Group | Number of Patients (N) | Number of Patients with<br>Therapeutic Cure (n) | Proportion of Therapeutic Cure (%) | Difference (%) | P-value |
| Placebo | XXX | XXX | XX.X | | |
| Test | xxx | XXX | XX.X | XX.X | x.xxxx |
| Reference | XXX | XXX | XX.X | XX.X | X.XXXX |

The 90% confidence interval for the difference in proportions between test and reference was calculated using Yates' correction.

Superiority of Active treatments over Placebo were tested using a two-sided Cochran-Mantel-Haenszel (CMH) test, stratified by clinical site, at the 5% significance level using last observation carried forward (LOCF).

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX
#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

## T14.2.10 Summary of Analysis Results of Secondary Efficacy Endpoint Proportion of Patients in each Treatment Group Who are Considered a Clinical Cure at Day $56 \pm 4$

| <b>Equivalence:</b> | Per-Protocol Pop | oulation | | | |
|---|---|---|---|---|---|
| | | | | <b>Difference Between Treatments</b> | |
| Treatment<br>Group | Number of Patients (N) | Number of Patients with<br>Clinical Cure (n) | Proportion of Clinical Cure (%) | Difference (%) | 90% CI Evaluation |
| Test | xxx | XXX | XX.X | | |
| Reference | xxx | xxx | XX.X | xx.x | xx.x - xx.x |

#### **Superiority: modified Intent-to-Treat Population**

| | | | | Treatment vs. Placebo | |
|---|---|---|---|---|---|
| Treatment<br>Group | Number of Patients (N) | Number of Patients with<br>Clinical Cure (n) | Proportion of Clinical Cure (%) | Difference (%) | P-value |
| Placebo | xxx | XXX | XX.X | | |
| Test | XXX | XXX | XX.X | XX.X | x.xxxx |
| Reference | xxx | XXX | XX.X | XX.X | X.XXXX |

The 90% confidence interval for the difference in proportions between test and reference was calculated using Yates' correction.

Superiority of Active treatments over Placebo were tested using a two-sided Cochran-Mantel-Haenszel (CMH) test, stratified by clinical site, at the 5% significance level using last observation carried forward (LOCF).

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

## T14.2.11 Summary of Analysis Results of Secondary Efficacy Endpoint Proportion of Patients in each Treatment Group Who are Considered a Mycological Cure at Day $56\pm4$

| | | | _ | <b>Difference Between Treatments</b> | |
|---|---|---|---|---|---|
| Treatment<br>Group | Number of Patients (N) | Number of Patients with<br>Mycological Cure (n) | Proportion of Mycological Cure (%) | Difference (%) | 90% CI Evaluation |
| Test | XXX | XXX | XX.X | | |
| Reference | XXX | XXX | XX.X | xx.x | xx.x - xx.x |

#### **Superiority: modified Intent-to-Treat Population**

| | | | _ | Treatment vs. Placebo | |
|---|---|---|---|---|---|
| Treatment<br>Group | Number of Patients (N) | Number of Patients with<br>Mycological Cure (n) | Proportion of Mycological Cure (%) | Difference (%) | P-value |
| Placebo | XXX | XXX | XX.X | | |
| Test | XXX | XXX | XX.X | XX.X | x.xxxx |
| Reference | XXX | XXX | XX.X | XX.X | X.XXXX |

The 90% confidence interval for the difference in proportions between test and reference was calculated using Yates' correction.

Superiority of Active treatments over Placebo were tested using a two-sided Cochran-Mantel-Haenszel (CMH) test, stratified by clinical site, at the 5% significance level using last observation carried forward (LOCF).

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX

**Ketoconazole Cream 2%** 

Protocol / Study No. 71875502

## T14.3.1 Overall Summary of Adverse Events (Safety Population)

| Description | Test<br>(N = xxx)<br>n (%) | Reference<br>(N = xxx)<br>n (%) | Placebo<br>(N = xxx)<br>n (%) | Total<br>(N = xxx)<br>n (%) |
|---|---|---|---|---|
| Patients in Safety Analysis population | XXX | XXX | XXX | XXX |
| Patients with at least one AE | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) |
| Discontinued study product due to above AE | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx(xx.x) |
| AEs reported | Xxx | xxx | xxx | xxx |
| Mild | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Moderate | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Severe | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Not Related | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Related | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Death | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Serious AE | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

MedDRA Version 21.0

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX

**Ketoconazole Cream 2%** 

Protocol / Study No. 71875502

# T14.3.2 Summary of Frequency of Adverse Events by Body System (Safety Population)

| - | | | Γest<br>= xxx | _ | ference<br>= xxx | | acebo<br>= xxx | Overall | Fisher's<br>P-value |
|---|---|---|---|---|---|---|---|---|---|
| <b>Body System</b> | Preferred Term | Events | Patients<br>n (%) | Events | Patients<br>n (%) | Events | Patients<br>n (%) | Fisher's<br>P-value | Test vs.<br>Reference |
| Patients with at least one AE | Total | XX | xxx (xx.x) | XX | xxx (xx.x) | XX | xxx (xx.x) | 0.1234 | NA |
| Ear and labyrinth disorders | Ear pain etc. | XX | xxx (xx.x) | XX | xxx (xx.x) | XX | xxx (xx.x) | 0.0425 | 0.0372 |

etc.

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

N = number of patients in safety population in that particular group; n= number of patients with data available for that particular group; total % is based on N

MedDRA Version 21.0

Note to programmer: If the global Fisher's exact test is statistically significant among the three treatment groups at the 5% alpha level (i.e. p < 0.05), then Fisher's exact test using only the test and reference groups will be performed to identify any potential statistically significant differences that are clinically relevant between the two active treatment groups.

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX

**Ketoconazole Cream 2%** 

Protocol / Study No. 71875502

# T14.3.3 Summary of Frequency of Adverse Events by Relationship (Safety Population)

| | | Test<br># of Events<br>(N = xxx) | | # of 1 | Reference<br># of Events<br>(N = xxx) | | Placebo<br># of Events<br>(N = xxx) |
|---|---|---|---|---|---|---|---|
| <b>Body System</b> | MedDRA Term | Related<br>n (%) | Not Related<br>n (%) | Related<br>n (%) | Not Related<br>n (%) | Related<br>n (%) | Not Related<br>n (%) |
| Total AEs<br>Ear and labyrinth | Total | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| disorders | Ear pain Hypoacusis | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

N = Total number of events in that particular group; Percentage is based on total number of events.

MedDRA Version 21.0

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX

**Ketoconazole Cream 2%** 

Protocol / Study No. 71875502

# T14.3.4 Summary of Frequency of Adverse Events by Severity (Safety Population)

| | | Test<br># of Events<br>(N = xxx) | | | # of Events # of Events | | | | Placebo<br># of Events<br>(N = xxx) | |
|---|---|---|---|---|---|---|---|---|---|---|
| Body<br>System | MedDRA<br>Term | Mild<br>n (%) | Moderate<br>n (%) | Severe<br>n (%) | Mild<br>n (%) | Moderate<br>n (%) | Severe<br>n (%) | Mild<br>n (%) | Moderate<br>n (%) | Severe<br>n (%) |
| Total AEs<br>Ear and | Total | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| labyrinth disorders | Ear pain | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Hypoacusis | xx (xx.x) | xx(xx.x) | xx (xx.x) | xx (xx.x) | xx(xx.x) | xx(xx.x) | xx (xx.x) | xx(xx.x) | xx (xx.x) |

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

N = Total number of events in that particular group; Percentage is based on total number of events.

MedDRA Version 21.0

02/28/2019

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

**Ketoconazole Cream 2%** 

Protocol / Study No. 71875502

## T14.3.5 Summary of Frequency of Serious Adverse Events (Safety Population)

| Body System | Preferred <b>Term</b> | Test<br># Events | Reference<br># Events | Reference<br># Events |
|---|---|---|---|---|
| Injury, poisoning and procedural complications | Alcohol poisoning | XXX | XXX | XXX |

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

MedDRA Version 21.0

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

**Ketoconazole Cream 2%** 

Protocol / Study No. 71875502

## T14.3.6 Summary of Vital Signs (Safety Population)

| Vital Signs | Visit | Statistic | Test N = xxx | Reference<br>N = xxx | Placebo<br>N = xxx |
|---|---|---|---|---|---|
| Systolic Blood Pressure (mmHg) | Visit 1 | $\begin{matrix} n \\ Mean \pm SD \end{matrix}$ | $\begin{array}{c} xxx \\ xxx.x \pm xx.x \end{array}$ | $\begin{array}{c} xxx \\ xxx.x \pm xx.x \end{array}$ | $\begin{array}{c} xxx \\ xxx.x \pm xx.x \end{array}$ |
| | | Median<br>Range | xxx.x $xxx.x - xxx.x$ | XXX.X $XXX.X - XXX.X$ | XXX.X $XXX.X - XXX.X$ |

Visit 2

Visit 3/Early Termination

Diastolic Blood Pressure (mmHg) Pulse Rate (beats/min) Respiration Rate (breaths/min) Temperature (F)

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

N = Total number of events in that particular group; Percentage is based on total number of events.

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

## L16.2.1 Listing of Discontinued Patients

| Treatment<br>Group | Patient<br>Screening<br>Number | Patient<br>Randomization<br>Number | Discontinuation<br>Reason | Population |
|---|---|---|---|---|
| Test | XX-XXX | XXXX | Withdrawal by Patient | Per-Protocol |
| | XX-XXX | XXXX | Lost to Follow-up | Safety |

Reference Placebo

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502


OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX

## L16.2.2 Listing of Protocol Deviations

| Treatment<br>Group | Patient<br>Screening<br>Number | Patient<br>Randomization<br>Number | Event Description | Population | Significant<br>Protocol<br>Deviation |
|---|---|---|---|---|---|
| Test | XX-XXX | XXXX | Outside Visit Window (Visit 3) | Safety | No |

Reference Placebo

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

#### L16.2.3.1 Listing of Patients Excluded from the Per-Protocol Population

| Treatment<br>Group | Patient<br>Screening<br>Number | Patient<br>Randomization<br>Number | Exclusion Reason |
|---|---|---|---|
| Test | XX-XXX | XXXX | Significant protocol deviation |

Reference Placebo

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX Page 1 of N

L16.2.3.2 Listing of Patients Excluded from the modified Intent-to-Treat Population

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

## L16.2.4.1 Listing of Demographic Data

| Treatment<br>Group | Patient<br>Screening<br>Number | Patient<br>Randomization<br>Number | Age | Sex | Ethnicity | Race | Birth<br>Control |
|---|---|---|---|---|---|---|---|
| Test | xx-xxx | XXXX | 30 | Female | Not Hispanic or Latino | Black or African American | Double Barrier |

Reference Placebo

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX Created on: ddmmmyy hh:mm Page 1 of N

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX

## L16.2.4.2 Listing of Medical History

| Treatment<br>Group | Patient<br>Screening<br>Number | Patient<br>Randomizatio<br>Number | n System | Diagnosis or<br>Surgical<br>Procedure | Start Date | End Date | Ongoing | Number of Tinea Pedis infections in the past 12 months |
|---|---|---|---|---|---|---|---|---|
| Test | XX-XXX | XXXX | Gynecologic | Menopause | //2012 | mm/dd/yyyy | | XXX |

Reference Placebo

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

#### L16.2.4.3 Listing of Prior and Concomitant Medication

| Treatment<br>Group | Patient<br>Screening<br>Number | Patient<br>Randomization<br>Number | Treatment<br>Area | Medication | Dosage/Unit | Frequency* | Route | Start/End<br>Date/ Ongoing | Indication | Prior? |
|---|---|---|---|---|---|---|---|---|---|---|
| Test | xx-xxx | XXXX | No | Lisinopril | 20 MG | QD | PO | //2017/<br>08/12/2017 | Hypertension | No |

Reference Placebo

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

\*PRN - As needed; QD - Daily (once per day); Q4H - Every 4 hours; Q8H - Every 8 hours; Q12H - Every 12 hours; BID - Twice per day; TID - 3

times per day; QID - 4 times per day; QOD - Every other day; QS - Every week; QM - Every month; Q3M - Every 3 months

 $PROGRAM: L: \DEV\755\71875502\SAS\PGM\XXXX$ 

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX

## L16.2.5 Listing of Drug Administration

| Treatment<br>Group | Patient<br>Screening<br>Number | Patient<br>Randomization<br>Number | Date of<br>First Dose | Date of<br>Last Dose | Total Doses<br>Applied | Missed<br>Doses | Treatment<br>Compliance |
|---|---|---|---|---|---|---|---|
| Test | XX-XXX | XXXX | mm/dd/yyyy | mm/dd/yyyy | XX | XX | Yes |

Reference Placebo

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

## **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX

## L16.2.6.1 Listing of Local Signs and Symptoms

| Treatment<br>Group | Patient<br>Screening<br>Number | Patient<br>Randomi<br>-zation<br>Number | Visit | Evaluator | Erythema | Scaling | Pruritus | | Maceration | | Total<br>Severity<br>Score | Clinical<br>Cure/<br>Failure |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Test | XX-XXX | XXXX | 1 | XXX | 0 | 0 | 0 | 1 | 0 | 0 | 1 | _ |
| | | | 2 | XXX | 0 | 0 | 0 | 1 | 0 | 0 | 1 | |
| | | | 3 | XXX | 0 | 0 | 0 | 1 | 0 | 0 | 1 | Cure |

Reference Placebo

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

## L16.2.6.2 Listing of Mycological Culture and KOH Wet Mount Results

| Treatment<br>Group | Patient<br>Screening<br>Number | Patient<br>Randomization<br>Number | Visit | Mycological<br>Culture | KOH<br>Wet Mount | Mycological<br>Cure/Failure | Therapeutic<br>Cure/Failure |
|---|---|---|---|---|---|---|---|
| Test | xx-xxx | XXXX | 1 | T. rubrum/E. floccosum | Positive | | |
| | | | 2 | T. rubrum/E. floccosum | Negative | | |
| | | | 3 | Negative | Negative | Cure | Cure |
| | | xx-xxxx | 1 | T. rubrum | Positive | | |
| | | | 2 | T. rubrum | Negative | | |
| | | | 3 | T. rubrum | Negative | Failure | Failure |
| Reference<br>Placebo | | | | | | | |

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

## L16.2.7.1 Listing of Treatment Emergent Adverse Events by Treatment

| Treatment<br>Group | Patient<br>Screening<br>Number | Patient<br>Randomi-<br>zation<br>Number | Body System /<br>MedDRA Term /<br>AE Term | Treatment<br>Area | Start /End<br>Date/<br>Ongoing | Severity | Relationship<br>to Study<br>Drug | Outcome | Action Taken/<br>Other Action<br>Taken | SAE |
|---|---|---|---|---|---|---|---|---|---|---|
| Test | xx-xxx | XXXX | Nervous system disorders /<br>Headache /<br>Headache | No | mm/dd/yyyy /<br>mm/dd/yyyy | Mild | Related | Recovered | Dose Not<br>Changed/<br>None | No |

Reference Placebo

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

## **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

## L16.2.7.2 Listing of Pre-treatment Adverse Events

| Patient<br>Screening<br>Number | Patient<br>Randomi-<br>zation<br>Number | Body System /<br>MedDRA Term /<br>AE Term | Treatment<br>Area | Start /End<br>Date/<br>Ongoing | Severity | Relationship<br>to Study<br>Drug | Outcome | Action Taken/<br>Other Action<br>Taken | SAE |
|---|---|---|---|---|---|---|---|---|---|
| XX-XXX | XXXX | Nervous system disorders / | No | mm/dd/yyyy / | Mild | Related | Recovered | Dose Not | No |
| | | Headache / | | mm/dd/yyyy | | | | Changed/ | |
| | | Headache | | | | | | None | |

 $PROGRAM: L: \DEV\755\71875502\SAS\PGM\XXXX$ 

Created on: ddmmmyy hh:mm

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

## L16.2.8.1 Listing of Pregnancy Test Results

| Treatment<br>Group | Patient<br>Screening<br>Number | Patient<br>Randomization<br>Number | Visit 1 | Visit 2 | Visit 3 /<br>Early Termination |
|---|---|---|---|---|---|
| Test | XX-XXX | XXXX | Negative | Negative | Negative |

Reference Placebo

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX

#### **Ketoconazole Cream 2%**

Protocol / Study No. 71875502

## L16.2.8.2 Listing of Vital Signs

| Treatment<br>Group | Patient<br>Screening<br>Number | Patient<br>Randomization<br>Number | Visit | Systolic BP (mmHg) | Diastolic BP<br>(mmHg) | Pulse Rate<br>(beats/min) | Respiration<br>Rate<br>(breaths/min) | Temperature<br>(F) |
|---|---|---|---|---|---|---|---|---|
| Test | XX-XXX | XXXX | Visit 1 | 120 | 70 | 84 | 18 | 98.6 |
| | | | Visit 2 | 140 | 100 | 74 | 18 | 97.0 |
| | | | Visit 3 | 140 | 100 | 74 | 18 | 97.0 |

Reference Placebo

Test: Ketoconazole Cream 2% (Encube Ethicals Pvt Ltd)

Reference: Ketoconazole Cream 2% (G&W Laboratories Inc.; Registrant: Teva Pharmaceuticals USA Inc.)

Placebo: Placebo Cream (Test vehicle) (Encube Ethicals Pvt Ltd)

PROGRAM: L:\DEV\755\71875502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71875502\SAS\OUT\XXXX